CLINICAL TRIAL: NCT02625532
Title: Early Follicular Phase vs Lutheal Phase Ovarian Stimulation in Bologna Criteria IVF/ICSI Cycles: A Randomized Comparative Single Center Trial. LUTEAL Trial
Brief Title: Early Follicular Phase vs Lutheal Phase Ovarian Stimulation in Bologna Criteria IVF/ICSI Cycles (LUTEAL Trial)
Acronym: LUTEAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto Bernabeu (Other)
Responsible Party: Principal Investigator, Joaquín Llácer, Gynaecologist. Reproductive Medicine Specialist at Instituto Bernabeu, Instituto Bernabeu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BER-LUT-2015-02; 2015-003856-31 (EudraCT Number)
Record Dates: First submitted 2015-11-09; First posted 2015-12-09 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Reproductive Techniques, Assisted
Keywords: Controlled Ovarian stimulation; Follicular phase; Luteal phase; Reproductive Techniques, Assisted
MeSH Terms: conditions — Helping Behavior | interventions — Follicular Phase; Luteal Phase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Follicular phase (Active Comparator): Controlled ovarian stimulation starts during follicular phase on day 2-3 of the menstrual cycle
  Interventions: Procedure: Follicular phase
- Luteal phase (Experimental): Controlled ovarian stimulation starts during luteal phase on day 3 to 5 after first LH positive urine test
  Interventions: Procedure: Luteal phase

INTERVENTIONS:
Procedure: Follicular phase — Controlled ovarian stimulation starts on day 2-3 of the menstrual cycle with recombinant recombinant FSH + LH, adding cetrorelix when the follicles reach 14 mm size and ovarian maturation with triptorelin acetate
  Other Names: Ovarian stimulation starts during the follicular phase
  Arms: Follicular phase
Procedure: Luteal phase — Controlled ovarian stimulation is started between 3rd and 5th day after the first LH positive urine test, adding cetrorelix when follicles reached 14 mm size and ovarian maturation with triptorelin acetate
  Other Names: Ovarian stimulation starts during the luteal phase
  Arms: Luteal phase

SUMMARY:
Exploratory, prospective, randomized, comparative, open trial with control group treated to assess the efficacy of follicular phase ovarian stimulation compared to lutheal phase ovarian stimulation in women with Bologna criteria for poor ovarian response.

DETAILED DESCRIPTION:
Two arms is established, the study group that will start ovarian stimulation in the luteal phase and the control group that will start ovarian stimulation in the follicular phase.

The randomization will be made in the 2-3 day of the menstrual cycle, according to a list of random allocation of treatments. After check that there is no contraindication to start the stimulation, the patients will be assigned to the treatment group.

The patients in the control group (follicular phase group) will start stimulation with two vials of 150 IU recombinant FSH + 75 IU recombinant LH (Pergoveris® 150/75). The patients in the study group (luteal phase group) will perform daily urine LH test from day 7th of the cycle and will start the administration of 150 IU recombinant FSH + 75 IU recombinant LH (Pergoveris® 150/75) at two vials daily from the 4th day of the LH positive test.

Antagonist cetrorelix acetate (Cetrotide® ) administration will start when the largest follicle shall be equal or greater than 14 mm. From this moment controls every 24-72 hours with foliculometría by ultrasound and blood hormone analysis with determination of estradiol and progesterone. For the final oocyte maturation 2 vials daily of 0.2 mg triptorelin acetate (Decapeptyl®) is administered. Oocyte collection will be made by transvaginal ultrasound-guided puncture according to IB protocol

The dosages and protocols used will be the usual for patients with diagnostic of poor ovarian response.

ELIGIBILITY:
Inclusion Criteria:

* Patient Bologna meets the criteria to be diagnosed as low responder
* Age under 41 years
* Regular menstrual cycles between 21 and 35 days
* Indication of in vitro fertilization
* Indication of start stimulation with 300 IU of FSH
* Presence of both ovaries
* Ability to participate and comply with the study protocol
* Having signed the written consent form

Exclusion Criteria:

* Presence of follicles larger than 10 mm in the randomization visit
* Endometriosis III / IV
* Concomitant uterine pathology: adenomyosis, submucosal myomas, Asherman's syndrome...
* Concurrent participation in another study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
number of oocytes in metaphase II obtained | Through study completion, average 2 weeks
  number of oocytes in metaphase II obtained by follicular puncture

SECONDARY OUTCOMES:
number of oocytes cumulus complexes | Through study completion, average 2 weeks
  number of oocytes cumulus complexes obtained by follicular puncture
duration of stimulation (days) | Through study completion, average 2 weeks
  number of days from the start of ovarian stimulation until the day of follicular puncture
cycle cancellation rate | Through study completion, average 2 weeks
  ratio of canceled cycles regarding the number of ovarian stimulation cycles initiated
Luteinizing hormone levels following administration of agonist for final oocyte maturation | Through study completion, average 2 weeks
  Luteinizing hormone blood levels the day after administration of agonist for final oocyte maturation
occurrence of side effects | Through study completion, average 2 weeks
  occurrence of side effects at the end of study
fertilization rate | Through study completion, average 2 weeks
  Number of correct fertilization oocytes 18 hours post-insemination

CONTACTS AND LOCATIONS:
Overall Officials: Joaquín Llácer, Principal Investigator — Instituto Bernabeu
Locations (1):
- Instituto Bernabeu, Alicante, Spain

REFERENCES:
- [Derived] Llacer J, Moliner B, Luque L, Bernabeu A, Lledo B, Castillo JC, Guerrero J, Ten J, Bernabeu R. Luteal phase stimulation versus follicular phase stimulation in poor ovarian responders: results of a randomized controlled trial. Reprod Biol Endocrinol. 2020 Feb 7;18(1):9. doi: 10.1186/s12958-020-00570-7. PMID 32033610